CLINICAL TRIAL: NCT02265185
Title: Measuring the Weight Status, Primary Care Usage and Dietary Intake in the Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1409-091
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED Patients: Children aged 2-10 visiting the Emergency Department.

SUMMARY:
Childhood obesity is a major area of concern for health care and public health. Overweight children are more likely overweight and obese adults. Chronic health problems associated with adult obesity are now occurring more frequently in children. Because of the associated health problems and potential for long term struggles with obesity, intervention early in life is essential for addressing the obesity epidemic. Some intervention work in this area has focused on the pediatric primary care setting in order to utilize the influence and credibility of medical providers. Unfortunately, primary care visits are often too short to spend a significant amount of time on issues of diet, weight and nutrition.

There has been very little work exploring the potential of alternative care settings, such as the pediatric Emergency Department (ED) in addressing childhood obesity. While provider time is also limited in the ED, there is often a considerable amount of downtime during emergency department visits that could be valuable time for patient and parent education. There may also be an opportunity to reach parents and children in the ED who do not regularly utilize primary care. In order to explore the possibility of pediatric obesity interventions in Children's Pediatric Emergency Department, we will need to measure the prevalence of obesity in the population that utilizes the Children's ED. The height of patients seen in the ED is not routinely measured, which makes calculating BMI to determine obesity impossible. This study, establishing the prevalence of obesity in Children's Emergency Department will lay the groundwork for future work addressing obesity in the ED.

DETAILED DESCRIPTION:
Background/Significance Childhood obesity is a well-documented public health crisis. Data from the most recent National Health and Nutrition Examination survey (NHANES) indicate that the prevalence of obesity is 8.4% in 2 to 5-year-olds, 17.7% in 6 to 11-year-olds, and 20.5% in 12 to 19-year-olds (1). Large racial/ethnic disparities in risk for obesity are already present by the preschool years (2). In 2 to 5-year-olds, 3.5% of non-Hispanic white children are obese, compared to 11.3% of non-Hispanic black and 16.7% of Hispanic children (1). Many health problems that were previously associated only with adult obesity are now being seen in youth, including the metabolic syndrome, type 2 diabetes, and cardiovascular abnormalities (3). Obesity tracks into adulthood, highlighting the need for early intervention (4). Overweight children have more chronic conditions, a greater risk of emergency department visits, and significantly higher costs for common pediatric hospitalizations (5-7). Successfully addressing the childhood obesity epidemic will require coordinated and collective efforts across many settings including multiple healthcare settings (8). Obesity interventions are increasingly being developed that utilize the influential role and credibility of pediatric primary care providers by integrating interventions into healthcare settings (9). Unfortunately, primary care visits are often short (average primary visit is 16.4 minutes) and leave little time for addressing obesity in detail, highlighting the need to also incorporate assessment and treatment in alternative care settings (i.e., emergency care) (10, 11).

There is little research on what role alternative healthcare setting could play in addressing childhood obesity. The pediatric ED is currently untapped as a setting for obesity screening, treatment and prevention (12). Yet, childhood obesity has important implications for emergency medicine and trauma care, and the pediatric ED may be shouldering a disproportionate burden of this disease compared to other healthcare settings (13, 14). Not addressing a patient's obesity in the ED setting is a missed opportunity, especially when many visits are obesity- related (e.g., asthma, type 2 diabetes, fractures), and weight reduction in specific subgroups could lead to a decrease in future ED utilization. The pediatric ED may not seem like an ideal location for addressing childhood obesity but many visits are for non-emergent/urgent conditions and these types of visits provide a window for screening and intervention (12,15). Families spend a substantial amount of time in the ED waiting for laboratory/radiology results and disposition. In 2013, the average length of stay in the Children's EDs was 155 minutes in Minneapolis and 143 minutes in St. Paul, valuable time that could be used for obesity screening, education, and connection to external resources. The pediatric ED has the potential to be an important additional healthcare setting for obesity screening, education, and linkage to external resources, but much more research is needed (12,13,16).

Three previous studies have examined obesity rates in the pediatric ED, each finding a higher prevalence of obesity compared to the general population (12,13,16). Prendergast et al. conducted a retrospective chart review and found a prevalence of obesity of 29% in a Chicago pediatric ED, nearly double the national average of 17% (12). The other two studies collected cross-sectional data from small samples in urban pediatric EDs and found a prevalence of obesity of 24% (13) and 21.6% (16). Only one study has tested obesity screening in the pediatric ED (16). Vaughn et al. found that all parents were receptive to obesity screening and prevention in the ED, regardless of race (16). They also found that only 7.6% of parents reported that their child's regular physician had counseled them regarding their child's weight, highlighting the need for obesity screening in additional healthcare settings (16). These studies indicate that pediatric EDs are seeing a population of patients at high risk for obesity, many of whom may not be receiving screening or counseling from their regular physician. Other topics in emergency medicine have received far greater coverage in the literature, including smoking cessation, injury prevention and substance abuse (13). With the dramatic increase in pediatric obesity, research on obesity in the pediatric ED is especially warranted as innovative strategies and collaboration across healthcare settings will be needed to successfully address this epidemic.

Currently, the prevalence of obesity in patients who utilize the pediatric ED at Children's Hospitals and Clinics of Minnesota is unknown. Because of time constraints, the height of patients seen in the pediatric ED are not routinely measured or recorded in the Electronic Medical Record (EMR). Establishing prevalence of obesity in this population is not possible without measuring the height of PED patients to determine BMI. Establishing the prevalence in the population of patients who utilize the pediatric ED will lay the groundwork for future grant proposals and research in this area.

Research Questions:

1. What is the prevalence of obesity in the Children's ED patient population?
2. What is the association between weight status and ED utilization for injury, asthma and mental health?

Study Design We will conduct a cross-sectional cohort study of patients aged 2-10 in Children's ED.

Methods ED research assistants will screen the ED log for patients in the 2-10 age range triaged level 3-5. Research assistants will randomly determine 1 out of 5 patients to approach for study enrollment. After the consent process is completed, the research assistant will measure and record the child's height, and ask the parent to complete a short questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Emergency Severity Index (ESI) Triage levels 3-5
2. Patient between 2 and 10 years of age (inclusive)
3. Parent able to consent

Exclusion Criteria:

1. Transferred patients

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients (aged 2-10) visiting the Children's EDs, who are triaged level 3-5, when a study RA is on duty will be eligible for the study. We have selected the 2-10 year old patient population for this study as the early grade school years are a critical time to intervene before unhealthy lifestyle habits are established, and this age group provides a unique window of opportunity in which to utilize parent and child interaction.
Sampling Method: Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Obesity | 1 year
  Prevalence in Children's ED will be compared to prevalence in the general pediatric population using previously established national data

SECONDARY OUTCOMES:
Associations between obesity and primary diagnosis | 1 year
  We will calculate attributable risk in the exposed population (in the obese) and attributable risk in the population (overall).

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Cutler, PhD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis and Saint Paul, Minnesota, United States